CLINICAL TRIAL: NCT00894569
Title: Open-Labeled, Randomized Multi-Center Phase II Study Evaluating the Efficacy and Safety of Paclitaxel/ Carboplatin With and Without Cetuximab as First-Line Treatment of Adeno- and Undifferentiated Carcinoma of Unknown Primary (CUP)
Brief Title: Paclitaxel/Carboplatin With or Without Cetuximab in CUP
Acronym: PACET-CUP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Prof. Dr. Alwin Krämer, University Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2008-003174-18
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Neoplasms, Unknown Primary; Carcinoma
Keywords: carcinoma of unknown primary; cancer of unknown primary; CUP; carboplatin; paclitaxel; cetuximab
MeSH Terms: conditions — Neoplasms, Unknown Primary; Carcinoma | interventions — CP protocol; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): 6 cycles of carboplatin/paclitaxel
  Interventions: Drug: paclitaxel/carboplatin
- B (Experimental): carboplatin/paclitaxel plus cetuximab until disease progression
  Interventions: Drug: paclitaxel/carboplatin; Drug: cetuximab

INTERVENTIONS:
Drug: paclitaxel/carboplatin — 6 cycles paclitaxel 175 mg/m² and carboplatin AUC 5, repetition d22.
Drug: cetuximab — cetuximab (400 mg/m² first dose, 250 mg/m² weekly) until disease progression
  Arms: B

SUMMARY:
The purpose of this study is to determine whether an addition of cetuximab to carboplatin/paclitaxel can improve efficacy in comparison to carboplatin/paclitaxel in patients with carcinoma of unknown-primary.

DETAILED DESCRIPTION:
Carcinomas of unknown primary (CUP) account for approximately 2-5% of all cancer diagnoses. Except for some subsets with favorable prognosis, for most of these patients, treatment options are limited, and no standard first-line regimen has been identified. Standard therapy for patients with adeno- or undifferentiated CUP is Paclitaxel/Carboplatin, yielding response rates between 20-40%. In recent years, targeted therapies with inhibitors to EGFR, several tyrosine kinases, and VEGF have been shown to improve survival in different solid tumor entities. Cetuximab, a monoclonal antibody against the EGF receptor, has proved efficacy in combination with chemotherapy in patients with metastatic colorectal cancer, gastric cancer, squamous cell carcinoma of head and neck and non-small cell lung cancer (NSCLC). Because of these promising results it seems to be reasonable to examine the impact of adding cetuximab to standard chemotherapy with paclitaxel and carboplatin in patients with CUP.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic proven, non-resectable carcinoma of unknown primary (adenocarcinoma or non-differentiated carcinoma)
* Measurable tumor lesion(s) according to RECIST criteria
* WHO PS 0 to 1
* Paclitaxel/Carboplatin with or without Cetuximab in Adeno- and Undifferentiated CUP (PACET-CUP)
* Signed written informed consent
* ≥ 18 years of age
* Effective contraception for both male and female subjects if the risk of conception exists
* Adequate bone marrow function:

  * Neutrophiles blood cell count (NBC) ≥ 1,5x109/L
  * Platelet count ≥ 100x109/L
  * Hemoglobin ≥ 5,00 mmol/L (8 g/dL)
* Adequate liver and renal function:

  * Bilirubin ≤ 1,5 x upper normal level (UNL) and not increasing more than 25% within the last 4 weeks
  * ASAT and ALAT ≤ 2,5 x UNL or in case of liver metastases ≤ 5 x UNL
  * Serum creatinine ≤ 1.5 x UNL

Exclusion Criteria:

* Previous exposure to epidermal growth factor receptor-targeting therapy
* Previous chemotherapy except adjuvant treatment with progression of disease documented > 6 months after end of adjuvant treatment
* Radiotherapy or major abdominal or thoracic surgery within the last 4 weeks before inclusion
* Concurrent chronic systemic immunotherapy, chemotherapy or hormone therapy
* Investigational agents or participation in clinical trials within 30 days before treatment start in this study
* Clinically relevant coronary disease or myocardial infarction within 12 months before study entry
* Possibility of a curative local treatment (surgery and/or radiotherapy)
* Women with axillary node metastasis as predominant tumor site
* Women with peritoneal carcinomatosis as predominant tumor site
* Men < 50 years old with retroperitoneal or mediastinal lymph node +/- lung metastases as predominant tumor site
* Identification of the primary or suspicion of a specific tumor entity by reference histopathology (i.e., Her-2 positive or hormone receptor positive tumors corresponding to breast cancer, CK7-negative/CK20- positive tumors with high probability for colorectal cancer)
* Peripheral neuropathy > CTC grade I
* Previous malignancy within the last 5 years (except history of basal cell carcinoma of skin or pre-invasive carcinoma of the cervix with adequate treatment)
* History of severe psychiatric illness
* Life expectancy less than six weeks
* Drug or alcohol abuse
* Known hypersensitivity reaction to any of the components of the study treatment
* Pregnancy (absence to be confirmed by β-hCG test) or lactation period
* Brain metastasis and/or leptomeningeal disease (known or suspected)
* Acute or sub-acute intestinal occlusion or inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
The rate of progression free survival at 8 months after randomization, defined as the proportion of patients alive with stable disease, partial or complete response, according to RECIST is the primary endpoint for the final analysis. | 8 months after randomization

SECONDARY OUTCOMES:
Efficacy: Response rate, Median progression free survival (PFS), Overall survival (OS) Toxicity | until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Alwin Kraemer, Prof. Dr., Principal Investigator — University of Heidelberg, Medic. Dep. V
Locations (1):
- University Hospital Heidelberg, Med. Dep. v, Heidelberg, Germany

REFERENCES:
- [Derived] Folprecht G, Trautmann K, Stein A, Huebner G, Stahl M, Kasper S, Kretzschmar A, Kohne CH, Grunwald V, Hofheinz RD, Schutte K, Loffler H, Bokemeyer C, Kramer A; Arbeitsgemeinschaft Internistische Onkologie (AIO) - CUP Group. Adding cetuximab to paclitaxel and carboplatin for first-line treatment of carcinoma of unknown primary (CUP): results of the Phase 2 AIO trial PACET-CUP. Br J Cancer. 2021 Feb;124(4):721-727. doi: 10.1038/s41416-020-01141-8. Epub 2020 Nov 25. PMID 33235314